CLINICAL TRIAL: NCT03171532
Title: Comparison of Clinical and Functional Outcomes at 2 Years of 4-strand Versus 5-strand Hamstring Autograft in Anterior Cruciate Ligament (ACL) Reconstruction: A Prospective Randomized Controlled Trial
Brief Title: Clinical and Functional Outcomes at 2 Years of 4-strand Versus 5-strand Hamstring Autograft in Anterior Cruciate Ligament Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015/00652
Record Dates: First submitted 2017-02-09; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-02

CONDITIONS: Physical Activity
Keywords: ACL
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 strand hamstring ACL reconstruction (Active Comparator): The hamstring tendons will be harvested by standard technique and the lengths of the Semitendinosus and Gracilis tendons will be measured after clearing all adherent muscle tissue. The ends will be prepared and folded in middle to prepare4-strand graft.
  Interventions: Procedure: Strands of Hamstring Autograft in ACL reconstruction
- 5 strand hamstring ACL reconstruction (Active Comparator): The hamstring tendons will be harvested by standard technique and the lengths of the Semitendinosus (ST) and Gracilis (GR) tendons will be measured after clearing all adherent muscle tissue. For 5-strand graft, minimum length of ST and GR in consideration would be 24 cm and 16 cm respectively. For 5-strand group the ST tendon will be be folded twice and sutured on itself to make a three strand graft and then GR tendon will be folded once along with it to make a final 5-strand graft.
  Interventions: Procedure: Strands of Hamstring Autograft in ACL reconstruction

INTERVENTIONS:
Procedure: Strands of Hamstring Autograft in ACL reconstruction — The femoral and tibial ends will be tubularised and the final graft diameter will be recorded after passing through sizing cylinders graduated in 0.5mm increments. The femoral and tibial tunnels will be drilled as per standard technique for single bundle ACL reconstruction via trans-portal or trans-tibial route and both ends fixed by interference screw with additional post on the tibial end.

SUMMARY:
This study aims to study differences in clinical and functional outcomes at 2 years based on hamstring graft size after single bundle anatomic ACL reconstruction using either 4-strand or 5-strand hamstring grafts. We also propose to study the characteristics of hamstring graft in our subset of patients in Asian population context.

DETAILED DESCRIPTION:
This will be a prospective, randomized interventional study conducted at the National University Hospital under University Orthopaedics and Hand surgery Cluster during the period of December 2015 to December 2018. Study participants: The study will include 80 patients with complete Anterior Cruciate Ligament (ACL) tear undergoing primary arthroscopic reconstruction with ipsilateral hamstring autograft after written informed consent to participate in the study.

The subjects will be divided into two groups A) 4-strand hamstring or B) 5-strand hamstring group by block randomization using an online randomization generator (http://www.graphpad.com/quickcalcs). All the subjects will undergo the procedure by otherwise identical technique performed by single surgeon. At 1 and 2 years functional and subjective outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Clinical and MRI confirmed complete ACL tear
3. Ipsilateral hamstring autograft
4. Concomitant meniscus injury requiring either meniscus repair or partial menisectomy
5. Concomitant chondral injury Grade 0,1,2 (International Cartilage Repair Society)
6. Regular scheduled follow up with adherence to prescribed rehab protocol

Exclusion Criteria:

1. Non consent
2. Paediatric patient; age less than 18 years
3. Partial or incomplete ACL tear
4. Revision ACL surgery
5. Hamstring allograft
6. Multi-ligament injury of the knee (ACL and/or Posterior Cruciate Ligament, Medial Collateral Ligament, Lateral Collateral Ligament, Postero Lateral Corner)
7. Past history of knee surgery
8. Contra-lateral ACL injury or other ligament injury
9. Chondral injury Grade 3,4 (International Cartilage Repair Society)
10. Intra-articular fracture (past or current)
11. Radiologically evident osteoarthritis changes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) Sport/Rec Score (Function in Sport and Recreation) change from baseline | Baseline, 1 year and 2 years post op
  Patient reported outcome

SECONDARY OUTCOMES:
Tegner-Lysholm Score change from baseline | Baseline, 1 year and 2 years post op
  Patient reported outcome
International Knee Documentation Committee (IKDC) Grade change from baseline | Baseline, 1 year and 2 years post op
  Patient reported outcome
KOOS Pain change from baseline | Baseline, 1 year and 2 years post op
  Patient reported outcome
KOOS Symptoms change from baseline | Baseline, 1 year and 2 years post op
  Patient reported outcome
KOOS Function in daily living (KOOS ADL) change from baseline | Baseline, 1 year and 2 years post op
  Patient reported outcome
KOOS Knee-related Quality of Life (KOOS QOL) change from baseline | Baseline, 1 year and 2 years post op
  Patient reported outcome

CONTACTS AND LOCATIONS:
Overall Officials: Lingaraj Krishna, FRCS (Orth), Principal Investigator — National University Health System
Locations (1):
- National University Health System, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No